CLINICAL TRIAL: NCT06030804
Title: Impact of Perioperative Dexmedetomidine on Long-term Survival in Older Patients After Cancer Surgery: a Multicenter Randomized Trial
Brief Title: Perioperative Dexmedetomidine and Long-term Survival After Cancer Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-227
Record Dates: First submitted 2023-09-03; First posted 2023-09-11 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Elderly; Cancer Surgery; Dexmedetomidine; Long-Term Survivors
Keywords: Older patients; Cancer surgery; Dexmedetomidine; Long-term survival
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): A loading dose of dexmedetomidine (0.6 μg/kg) will be administered over 10-15 minutes before anaesthesia induction, followed by a continuous infusion at a rate of 0.5 μg/kg/h till 1 hour before the end of surgery. Patient-controlled dexmedetomidine supplemented sufentanil analgesia will be provided after surgery: the formula contains a mixture of sufentanil (1.25 μg/ml) and dexmedetomidine (1.25 μg/ml), diluted with normal saline to a total volume of 160 ml; the analgesic pump is set to administer a background infusion at a rate of 1 ml/h, with patient-controlled bolus of 2 ml each time and a lockout time of 8 minutes.
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): Volume-matched normal saline will be administered in the same rate and volume for the same duration as in the dexmedetomidine group during anesthesia. Patient-controlled sufentanil analgesia will be provided after surgery: the formula contains sufentanil (1.25 μg/ml), diluted with normal saline to a total volume of 160 ml; the analgesic pump is set to administer a background infusion at a rate of 1 ml/h, with patient-controlled bolus of 2 ml each time and a lockout time of 8 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — A loading dose of dexmedetomidine (0.6 μg/kg) will be administered over 10-15 minutes before anaesthesia induction, followed by a continuous infusion at a rate of 0.5 μg/kg/hr till 1 hour before the end of surgery. Patient-controlled dexmedetomidine supplemented sufentanil analgesia will be provided after surgery: the formula contains a mixture of sufentanil (1.25 μg/ml) and dexmedetomidine (1.25 μg/ml), diluted with normal saline to a total volume of 160 ml; the analgesic pump is set to administer a background infusion at a rate of 1 ml/h, with patient-controlled bolus of 2 ml each time and a lockout time of 8 minutes.
  Other Names: Dexmedetomidine hydrochloride
  Arms: Dexmedetomidine group
Drug: Placebo — Volume-matched normal saline will be administered in the same rate and volume for the same duration as in the dexmedetomidine group during anesthesia. Patient-controlled sufentanil analgesia will be provided after surgery: the formula contains sufentanil (1.25 μg/ml), diluted with normal saline to a total volume of 160 ml; the analgesic pump is set to administer a background infusion at a rate of 1 ml/h, with patient-controlled bolus of 2 ml each time and a lockout time of 8 minutes.
  Other Names: Normal saline
  Arms: Control group

SUMMARY:
Along with aging population, cancer incidence and mortality are increasing. However, despite advances in oncology and surgery, long-term survival of cancer patients is far from optimal. Dexmedetomidine is a highly selective alpha 2 adrenergic receptor agonist with sedative, analgesic, and anxiolytic effects. Studies showed that perioperative use of dexmedetomidine reduces delirium and some non-delirium complications after surgery. In long-term follow-up studies of older patients who, for other reasons, were randomized to receive either dexmedetomidine or placebo during intra- or postoperative period, dexmedetomidine use was associated with improved long-term survival. This multicenter randomized trial aims to investigate the effect of perioperative dexmedetomidine on long-term outcomes in older patients undergoing cancer surgery.

DETAILED DESCRIPTION:
Along with aging population, cancer incidence and mortality are increasing. Surgical resection remains the mainstay treatment for solid organ cancer. However, despite advances in oncology and surgery, long-term survival of cancer patients is far from optimal. For example, the 5-year survival rate of cancer patients is about 36.9% in China, and the survival rate decreases for about 10% each year in older patients after cancer surgery. How to improve long-term survival after cancer surgery remains an urgent problem to be solved.

Cancer death usually occur after cancer recurrence or metastasis. The development of cancer recurrence or metastasise after surgical resection depends on the balance between the anti-cancer defense function of host and the invasiveness of residual cancer cells. Studies showed that surgery, while resecting cancer mass, also releases cancer cells into the circulation. Surgical stress also impairs cell-mediated immunity and promote cancer growth.

Dexmedetomidine is a highly selective alpha 2 adrenergic receptor agonist with sedative, analgesic, and anxiolytic effects. Studies showed that intraoperative use of dexmedetomidine reduces anesthetic and opioid consumption and relieves surgery-related stress response and inflammation. Studies also showed that perioperative use of dexmedetomidine reduces delirium, a commonly occurred complication in older patients, and some non-delirium complications after surgery.

The effect of perioperative dexmedetomidine on long-term outcomes after cancer surgery remains unclear. In a long-term follow-up of older patients who were randomized to receive either low-dose dexmedetomidine or placebo during intensive care unit stay, dexmedetomidine use was associated with improved survival within 2 years. In a recent long-term follow-up of older patients who were randomized to receive either dexmedetomidine or placebo during surgery, dexmedetomidine use was associated with improved recurrence-free survival.

The investigators hypothesize that perioperative use of dexmedetomidine may improve long-term survival after cancer surgery. This multicenter randomized trial aims to investigate the effect of perioperative dexmedetomidine on long-term outcomes in older patients undergoing cancer surgery.

ELIGIBILITY:
Inclusion criteria:

1. Aged 60 years or older.
2. Scheduled to undergo radical surgery for cancer under general anesthesia, with an expected surgical duration of 2 hours or longer.
3. Required patient-controlled intravenous analgesia after surgery.

Exclusion criteria:

1. Inability to communicate preoperatively due to visual, auditory, verbal. or other reasons.
2. Surgery for breast cancer or intracranial tumor.
3. Preoperative severe sinus bradycardia (<50 beats per minute), sick sinus syndrome，or second-degree or above atrioventricular block without pacemaker.
4. Severe hepatic dysfunction (Child-Pugh class C).
5. Severe renal dysfunction (requirement of renal replacement therapy before surgery).
6. Enrolled in other clinical studies.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4532 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival after surgery | Up to 3 years after surgery of the last enrolled patient.
  Time interval from index surgery to cancer recurrence/metastasis/progression or all-cause death, whichever comes first.

SECONDARY OUTCOMES:
Incidence of postoperative delirium. | During the first 4 postoperative days.
  Delirium will be assessed with the 3D-Confusion Assessment Method (3D-CAM) or CAM for the Intensive Care Unit (CAM-ICU) twice daily during the first 4 postoperative days.
Incidence of cognitive dysfunction at 6 months and 1 year postoperatively. | At 6 months and 1 year postoperatively.
  Cognitive function will be assessed with the Telephone Montreal Cognitive Assessment (T-MoCA; scores range from 0 to 22, with higher score indicating better function) before surgery and at 6 months and 12 months after surgery. A T-MoCA score reduction of 1 standard deviation (SD) or more from baseline will be considered occurrence of cognitive dysfunction.

OTHER OUTCOMES:
Rate of intensive care unit (ICU) admission after surgery. | Up to 30 days after surgery.
  Percentage of patients who required ICU admission within 30 days after surgery.
Intensity of pain after surgery. | Two hours after surgery and during the first 4 postoperative days.
  Intensity of pain will be assessed with the Numeric Rating Scale (NRS; an 11-point scale where 0=no pain and 10=the worst pain) twice daily during the first 4 postoperative days.
Subjective sleep quality after surgery. | During the first 4 postoperative days.
  Subjective sleep quality will be assessed with the Numeric Rating Scale (NRS; an 11-point scale where 0=the best sleep and 10=the worst sleep) once daily during the first 4 postoperative days.
Length of stay in hospital after surgery. | Up to 30 days after surgery.
  Length of stay in hospital after surgery.
Incidence of postoperative complications within 30 days. | Up to 30 days after surgery.
  Postoperative complications are defined as new-onset medical events other than delirium that are deemed harmful and require therapeutic intervention, that is grade II or higher on the Clavien-Dindo classification.
Overall survival after surgery | Up to 3 years after surgery of the last enrolled patient.
  Time interval from index surgery to all-cause death.
Cancer-specific survival after surgery | Up to 3 years after surgery of the last enrolled patient.
  Time interval from index surgery to cancer-specific death, with deaths from other causes being censored at the time of death. Cancer-specific death is defined as death fully attributable to the cancer for which the index surgery is performed and usually involves cancer recurrence/metastasis/progression after exclusion of other causes such as stroke and myocardial infarction.
Event-free survival after surgery | Up to 3 years after surgery of the last enrolled patient.
  Time interval from index surgery to cancer recurrence/metastasis/progression, new-onset cancer, new-onset serious illness (requiring hospitalization), or all-cause death, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD,PhD, Principal Investigator — Peking University First Hospital
Locations (39):
- China (39):
  - The First Affiliated Hospital of China University of Science and Technology, Hefei, Anhui
  - The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital), Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Tsinghua University Yuquan Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Army Medical University (Southwest Hospital), Chongqing, Chongqing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Jinjiang City Hospital (Shanghai Sixth People's Hospital, Fujian Hospital), Jinjiang, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Shenzhen University, Shenzhen, Guangdong
  - The Second Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Affiliated Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - Zhejiang Cancer Hospital, Zhejiang, Hangzhou
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tangshan Workers' Hospital, Tangshan, Hebei
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Xiangya Hospital Central South university, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Nanjing General Hospital of Nanjing Military Region, Nanjing, Jiangsu
  - Affiliated Drum Tower Hospital, Medical School of Nanjing University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - Bethune First Hospital Of Jilin University, Changchun, Jilin
  - General hospital of eastern theater command, Nanjing, Nanjing
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi
  - Shandong Provincial Hospital Heze Hospital, Heze, Shandong
  - Shanghai Fourth People's Hospital Affiliated to Tongji University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Zhang DF, Su X, Meng ZT, Li HL, Wang DX, Xue-Ying Li, Maze M, Ma D. Impact of Dexmedetomidine on Long-term Outcomes After Noncardiac Surgery in Elderly: 3-Year Follow-up of a Randomized Controlled Trial. Ann Surg. 2019 Aug;270(2):356-363. doi: 10.1097/SLA.0000000000002801. PMID 29742525
- [Background] Du YT, Li YW, Zhao BJ, Guo XY, Feng Y, Zuo MZ, Fu C, Zhou WJ, Li HJ, Liu YF, Cheng T, Mu DL, Zeng Y, Liu PF, Li Y, An HY, Zhu SN, Li XY, Li HJ, Wu YF, Wang DX, Sessler DI; Peking University Clinical Research Program Study Group. Long-term Survival after Combined Epidural-General Anesthesia or General Anesthesia Alone: Follow-up of a Randomized Trial. Anesthesiology. 2021 Aug 1;135(2):233-245. doi: 10.1097/ALN.0000000000003835. PMID 34195784
- [Background] Fokas E, Engenhart-Cabillic R, Daniilidis K, Rose F, An HX. Metastasis: the seed and soil theory gains identity. Cancer Metastasis Rev. 2007 Dec;26(3-4):705-15. doi: 10.1007/s10555-007-9088-5. PMID 17786535
- [Background] Khuri SF, Henderson WG, DePalma RG, Mosca C, Healey NA, Kumbhani DJ; Participants in the VA National Surgical Quality Improvement Program. Determinants of long-term survival after major surgery and the adverse effect of postoperative complications. Ann Surg. 2005 Sep;242(3):326-41; discussion 341-3. doi: 10.1097/01.sla.0000179621.33268.83. PMID 16135919
- [Background] Sessler DI. Long-term consequences of anesthetic management. Anesthesiology. 2009 Jul;111(1):1-4. doi: 10.1097/ALN.0b013e3181a913e1. No abstract available. PMID 19512884
- [Background] Yamaguchi K, Takagi Y, Aoki S, Futamura M, Saji S. Significant detection of circulating cancer cells in the blood by reverse transcriptase-polymerase chain reaction during colorectal cancer resection. Ann Surg. 2000 Jul;232(1):58-65. doi: 10.1097/00000658-200007000-00009. PMID 10862196
- [Background] Page GG, Blakely WP, Ben-Eliyahu S. Evidence that postoperative pain is a mediator of the tumor-promoting effects of surgery in rats. Pain. 2001 Feb 1;90(1-2):191-9. doi: 10.1016/s0304-3959(00)00403-6. PMID 11166986
- [Background] Heaney A, Buggy DJ. Can anaesthetic and analgesic techniques affect cancer recurrence or metastasis? Br J Anaesth. 2012 Dec;109 Suppl 1:i17-i28. doi: 10.1093/bja/aes421. PMID 23242747
- [Background] Melamed R, Rosenne E, Shakhar K, Schwartz Y, Abudarham N, Ben-Eliyahu S. Marginating pulmonary-NK activity and resistance to experimental tumor metastasis: suppression by surgery and the prophylactic use of a beta-adrenergic antagonist and a prostaglandin synthesis inhibitor. Brain Behav Immun. 2005 Mar;19(2):114-26. doi: 10.1016/j.bbi.2004.07.004. PMID 15664784
- [Background] Alazawi W, Pirmadjid N, Lahiri R, Bhattacharya S. Inflammatory and Immune Responses to Surgery and Their Clinical Impact. Ann Surg. 2016 Jul;264(1):73-80. doi: 10.1097/SLA.0000000000001691. PMID 27275778
- [Background] Liu S, Yu X, Ye F, Jiang L. Can the systemic inflammation score be used to predict prognosis in gastric cancer patients undergoing surgery? A systematic review and meta-analysis. Front Surg. 2022 Sep 19;9:971326. doi: 10.3389/fsurg.2022.971326. eCollection 2022. PMID 36338660
- [Background] Shakhar G, Ben-Eliyahu S. Potential prophylactic measures against postoperative immunosuppression: could they reduce recurrence rates in oncological patients? Ann Surg Oncol. 2003 Oct;10(8):972-92. doi: 10.1245/aso.2003.02.007. PMID 14527919
- [Background] Payne CJ, Gibson SC, Bryce G, Jardine AG, Berry C, Kingsmore DB. B-type natriuretic peptide predicts long-term survival after major non-cardiac surgery. Br J Anaesth. 2011 Aug;107(2):144-9. doi: 10.1093/bja/aer119. Epub 2011 May 24. PMID 21610013
- [Background] Straatman J, Cuesta MA, de Lange-de Klerk ES, van der Peet DL. Long-Term Survival After Complications Following Major Abdominal Surgery. J Gastrointest Surg. 2016 May;20(5):1034-41. doi: 10.1007/s11605-016-3084-4. Epub 2016 Feb 8. PMID 26857591
- [Background] Vakkila J, Lotze MT. Inflammation and necrosis promote tumour growth. Nat Rev Immunol. 2004 Aug;4(8):641-8. doi: 10.1038/nri1415. No abstract available. PMID 15286730
- [Background] Abdel-Meguid ME. Dexmedetomidine as anesthetic adjunct for fast tracking and pain control in off-pump coronary artery bypass. Saudi J Anaesth. 2013 Jan;7(1):6-8. doi: 10.4103/1658-354X.109557. PMID 23717223
- [Background] Jalonen J, Hynynen M, Kuitunen A, Heikkila H, Perttila J, Salmenpera M, Valtonen M, Aantaa R, Kallio A. Dexmedetomidine as an anesthetic adjunct in coronary artery bypass grafting. Anesthesiology. 1997 Feb;86(2):331-45. doi: 10.1097/00000542-199702000-00009. PMID 9054252
- [Background] Li Y, Wang B, Zhang LL, He SF, Hu XW, Wong GT, Zhang Y. Dexmedetomidine Combined with General Anesthesia Provides Similar Intraoperative Stress Response Reduction When Compared with a Combined General and Epidural Anesthetic Technique. Anesth Analg. 2016 Apr;122(4):1202-10. doi: 10.1213/ANE.0000000000001165. PMID 26991622
- [Background] Wang XW, Cao JB, Lv BS, Mi WD, Wang ZQ, Zhang C, Wang HL, Xu Z. Effect of perioperative dexmedetomidine on the endocrine modulators of stress response: a meta-analysis. Clin Exp Pharmacol Physiol. 2015 Aug;42(8):828-36. doi: 10.1111/1440-1681.12431. PMID 26016707
- [Background] Li B, Li Y, Tian S, Wang H, Wu H, Zhang A, Gao C. Anti-inflammatory Effects of Perioperative Dexmedetomidine Administered as an Adjunct to General Anesthesia: A Meta-analysis. Sci Rep. 2015 Jul 21;5:12342. doi: 10.1038/srep12342. PMID 26196332
- [Background] Duan X, Coburn M, Rossaint R, Sanders RD, Waesberghe JV, Kowark A. Efficacy of perioperative dexmedetomidine on postoperative delirium: systematic review and meta-analysis with trial sequential analysis of randomised controlled trials. Br J Anaesth. 2018 Aug;121(2):384-397. doi: 10.1016/j.bja.2018.04.046. Epub 2018 Jun 22. PMID 30032877
- [Background] Kong H, Xu LM, Wang DX. Perioperative neurocognitive disorders: A narrative review focusing on diagnosis, prevention, and treatment. CNS Neurosci Ther. 2022 Aug;28(8):1147-1167. doi: 10.1111/cns.13873. Epub 2022 Jun 1. PMID 35652170
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Li CJ, Wang BJ, Mu DL, Hu J, Guo C, Li XY, Ma D, Wang DX. Randomized clinical trial of intraoperative dexmedetomidine to prevent delirium in the elderly undergoing major non-cardiac surgery. Br J Surg. 2020 Jan;107(2):e123-e132. doi: 10.1002/bjs.11354. PMID 31903588
- [Background] Cata JP, Singh V, Lee BM, Villarreal J, Mehran JR, Yu J, Gottumukkala V, Lavon H, Ben-Eliyahu S. Intraoperative use of dexmedetomidine is associated with decreased overall survival after lung cancer surgery. J Anaesthesiol Clin Pharmacol. 2017 Jul-Sep;33(3):317-323. doi: 10.4103/joacp.JOACP_299_16. PMID 29109628
- [Background] Lavon H, Matzner P, Benbenishty A, Sorski L, Rossene E, Haldar R, Elbaz E, Cata JP, Gottumukkala V, Ben-Eliyahu S. Dexmedetomidine promotes metastasis in rodent models of breast, lung, and colon cancers. Br J Anaesth. 2018 Jan;120(1):188-196. doi: 10.1016/j.bja.2017.11.004. Epub 2017 Nov 23. PMID 29397129
- [Background] Xing MW, Li CJ, Guo C, Wang BJ, Mu DL, Wang DX. Effect of intraoperative dexmedetomidine on long-term survival in older patients after major noncardiac surgery: 3-year follow-up of a randomized trial. J Clin Anesth. 2023 Jun;86:111068. doi: 10.1016/j.jclinane.2023.111068. Epub 2023 Feb 1. PMID 36736209
- [Background] Austin PC. An Introduction to Propensity Score Methods for Reducing the Effects of Confounding in Observational Studies. Multivariate Behav Res. 2011 May;46(3):399-424. doi: 10.1080/00273171.2011.568786. Epub 2011 Jun 8. PMID 21818162